CLINICAL TRIAL: NCT02837003
Title: 3-Month Discontinuation of Dual Antiplatelet Therapy After Ultimaster Sirolimus-Eluting Stent Implantation
Acronym: MODEL U-SES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Teikyo University (Other)
Responsible Party: Sponsor
Other Study IDs: MODEL U-SES
Record Dates: First submitted 2016-07-08; First posted 2016-07-19 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Artery Disease
Keywords: Drug-Eluting Stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; thienopyridine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Experimental: Aspirin: Aspirin treatment for 3 months after the Ultimaster sirolimus-eluting stent implantation.
  Interventions: Drug: Aspirin
- Experimental: Thienopyridine: Thienopyridine treatment for 3 months after the Ultimaster sirolimus-eluting Stent implantation.
  Interventions: Drug: Thienopyridine

INTERVENTIONS:
Drug: Aspirin — Discontinuation of aspirin at 3 months after the Ultimaster sirolimus-eluting stent implantation by the physician's discretion.
  Groups: Experimental: Aspirin
Drug: Thienopyridine — Discontinuation of thienopyridine at 3 months after the Ultimaster sirolimus-eluting stent implantation by the physician's discretion.
  Groups: Experimental: Thienopyridine

SUMMARY:
To evaluate safety of reduction of dual antiplatelet therapy period to three months after implantation of Ultimaster sirolimus-eluting stent (U-SES).

Additionally to investigate appropriateness of thienopyridine monotherapy with discontinuation of aspirin.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery lesion who received percutaneous coronary intervention using Ultimaster sirolimus-eluting stent.
* Patients considered appropriate to discontinue dual antiplatelet therapy at 3 months after stent implantation.
* Patients who have provided written informed consent.

Exclusion Criteria:

* Patients previously experienced stent thrombosis.
* Patients who are unable to clinical follow-up procedure specified in the protocal for the present study.
* Patients who are enrolled or planned to participate in another clinical trials of antiplatelet therapy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The present study consisted of the following two study arms: the 3-month DAPT arm, a new registry arm in which 1,500 patients are consecutively recruite at 72 medical institutions; and the Longer DAPT arm, a historical control arm that consisted of 1,123 patients at 58 medical institutions.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of all cause death in 12 months, myocardial infarction, stroke (ischemic and hemorrhagic), ARC definite/probable stent thrombosis and serious bleeding (BARC 3 or 5). | 12-month

SECONDARY OUTCOMES:
Composite endpoint of all cause death in 3 months, myocardial infarction, stroke (ischemic and hemorrhagic), ARC definite/probable stent thrombosis and serious bleeding (BARC 3 or 5). | 3-month
Major adverse cardiac event | 3-month
Major adverse cardiac event | 12-month
All cause death | 3-month
All cause death | 12-month
Cardiac death | 3-month
Cardiac death | 12-month
Myocardial infarction | 3-month
Myocardial infarction | 12-month
Stroke (ischemic and hemorrhagic) | 3-month
Stroke (ischemic and hemorrhagic) | 12-month
Target lesion revascularization | 3-month
Target lesion revascularization | 12-month
Target vessel revascularization | 3-month
Target vessel revascularization | 12-month
Readmission related to angina | 3-month
Readmission related to angina | 12-month
Stent thrombosis | 3-month
Stent thrombosis (ARC definition) | 12-month
Bleeding complications (BARC definition) | 3-month
Bleeding complications (BARC definition) | 12-month
Comparison of event rate by the type of antiplatelet agent | 12-month

CONTACTS AND LOCATIONS:
Overall Officials: Ken Kozuma, MD, PhD, Principal Investigator — Teikyo University Hospital
Locations (1):
- Teikyo University Hospital, Tokyo, Japan